CLINICAL TRIAL: NCT02231346
Title: Berodual® Respimat® 20/50 Microgram/Dose Solution for Inhalation: Assessment of Handling and Patient Satisfaction in Comparison to a Powder Inhaler
Brief Title: Postmarketing Surveillance Study to Assess Handling and Patient Satisfaction on Berodual® Respimat® Solution for Inhalation in Comparison to a Powder Inhaler in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 215.1366
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- chronic obstructive pulmonary disease patients
  Interventions: Drug: Berodual® Respimat® - inhaler

INTERVENTIONS:
Drug: Berodual® Respimat® - inhaler

SUMMARY:
New perceptions about handling and patient satisfaction of the everyday use of Berodual® Respimat® compared to a powder inhaler in patients with chronic obstructive lung disease (COLD). Moreover, further knowledge should be attained about the tolerability of Berodual® Respimat®

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged at least 18 years
* Patients who are suffering from symptoms of a chronic obstructive lung disease (COLD) can be included in the PMS. To reduce influences caused by the use of a variety of different powder inhaler, only patients who are already regularly using Diskus® powder inhaler should be included, as the Diskus® as well as the Berodual® Respimat® are multiple dose devices
* During the PMS the Diskus® therapy is to be continued

Exclusion Criteria:

* Patients who meet one or more of the general or specific contraindications mentioned in the Summary of Product Characteristics (SmPC) are excluded from the Postmarketing Surveillance (PMS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of chronic obstructive pulmonary disease recruited at pneumologists in practice
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2005-10; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 4 weeks
Number of patients who prematurely discontinued therapy with Berodual® Respimat® | up to 4 weeks

SECONDARY OUTCOMES:
Assessment of patient satisfaction with regard to handling of Berodual® Respimat® inhaler | up to 4 weeks
  by means of a patient satisfaction and preference questionnaire (PASAPQ)
Assessment of patient satisfaction with regard to handling of Diskus® inhaler | Baseline
  by means of patient satisfaction and preference questionnaire (PASAPQ)